CLINICAL TRIAL: NCT04238858
Title: Effects of Subtenon-injected Autologous Platelet-rich Plasma on Visual Functions in Eyes With Retinitis Pigmentosa
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-596-16
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Growth factors; Platelet rich plasma; Visual functions
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Prospective open-label, before-after-control group comparisions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Before application (Active Comparator): Forty-nine eyes belonging to 37 patients before injection aPRP.
  Interventions: Biological: Platelet rich plasma
- After application (No Intervention): Forty-nine eyes belonging to 37 patients after injection aPRP.
- Sham application (Sham Comparator): 11 patients before - after aPPP injection
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: Platelet rich plasma — blood is drawn from the patient's antecubital vein and inserted into four 3.0 ml vacutainer tubes that contain trisodium citrate. These four tubes were placed in a centrifuge machine, and centrifugation was carried out at 2500 rpm (580×g) for 8 min within a 30-min blood collection period. As a result of centrifugation, the plasma was separated in the vacutainer tubes from the remaining blood components. Three different layers formed in the tubes: red blood cells at the bottom, aPRP in the middle layer, and aPPP in the top layer. A total of 1.5 ml of the middle layer (which mainly contained platelets) was withdrawn by syringe, and it was immediately injected into the subtenon space of each eye.
  Arms: Before application; Sham application

SUMMARY:
Purpose One of the main reasons for apoptosis and dormant cell phases in degenerative retinal diseases such as retinitis pigmentosa (RP) is growth factor withdrawal in the cellular microenvironment. Growth factors and neurotrophins can significantly slow down retinal degeneration and cell death in animal models. One possible source of autologous growth factors is platelet-richplasma.The purpose of this study was to determine if subtenon injections of autologous platelet-rich plasma (aPRP) can have beneficial effects on visual function in RP patients by reactivating dormant photoreceptors.

DETAILED DESCRIPTION:
More than 240 genetic mutations are involved in inherited retinal dystrophies, which constitute an overlapping group of genetic and clinical heterogeneous disorders. Retinitis pigmentosa (RP) is a heterogeneous genetic disorder (autosomal dominant, autosomal recessive, X-linked, or sporadic cases from spontaneous mutations) characterized by the progressive devolution of the retina and affecting 1/3000- 8000 people worldwide. Symptoms include generally diminishing visual fields starting in the mid-periphery and advancing toward the fovea, ultimately leading to visual impairment and blindness with waxy-colored optic atrophy. RP is also described as rod-cone dystrophy because of the primary degeneration of rods along with secondary degeneration of cones, with photoreceptor rods appearing to be more affected than cones. Diseased photoreceptors face apoptosis,which results in reducing the thickness of the outer nuclear layer and the retinal pigment epithelium layer with abnormal pigmentary deposits. Although apoptosis and photoreceptor loss are common outcomes of all genetic types, their clinical features and progression are not homogeneous. It is currently known that while some photoreceptor cells do die, others appear to be in suspended animation . In the photoreceptor microenvironment,when growth factor (GF) levels or their receptor activities decrease over an extended period, apoptosis and cell death occur. The length of this period differs with each genetic type. The time during which there is a decrease in the effects of growth factors until cell death, the photoreceptors can be described as being in sleep mode, on standby, or in a dormant phase. In this phase, cone photoreceptors are alive, but they cannot function. GFs and neurotrophins, such as basic fibroblast growth factor (bFGF), neural growth factor (NGF), ciliary neurotrophic factor (CNTF), and brain-derived neurotrophic factor (BDNF), can significantly slow retinal degeneration and cell death in animal models. One possible source of autologous GFs is platelet-rich plasma (PRP). PRP is defined as a biological product that features platelet concentration; it is collected from centrifuged whole blood. Through the activation ofa reactivator (such as sodium chloride or citrate), accumulated platelets can secrete a large quantity of preparations rich in growth factors (PRGFs) via the release of intracellular α-granules. PRGFs are an aggregation of cytokines that include transforming growth factors (TGF-β), interleukine-6 (IL-6), BDNF, and vascular endothelial growth factors (VEGF). The strong restoring function of autologous PRP (aPRP) is based mainly on the trophic capacity of PRGFs . Currently, PRP is being tested as a therapeutic option in some clinical situations, for example in orthopedics, ophthalmology, and healing therapies. Some pre-clinical and clinical trials have addressed the use of PRP and various GFs, such as the intravitreal injection of bFGF in retinal dystrophy and the topical applications of NGF to treat glaucoma and neurotrophic keratitis. The use of PRGFs in ophthalmology has been successfully applied to ocular surface disorders, including the treatment of ocular surface syndrome and flap necrosis after LASIK surgery. A recent study observed that administration of platelet-derived proteins adjacent to the lacrimal gland restored lacrimal function in all patients. The clinical and pre-clinical use of aPRP in ophthalmology has encouraged practitioners to use it through subtenon injection in the treatment of retinal diseases. Through the subtenon injection of PRP, the level of neurotrophic growth factors may be increased in the microenvironment around the photoreceptors, thus potentially reactivating photoreceptors that are in sleep mode.Fetal bovine serum,allogeneic serum,and umbilical cord serum have also been used as sources of growth factors, but they are heterologous products with a higher risk of allergic reactions and infectious disease transmission. In order to avoid these issues, and because of the accessibility and relatively safe nature of aPRP, we chose to use aPRP as a source of growth factors in our study. The purpose of this prospective open-label clinical trial was to determine whether the subtenon injection of aPRP may have beneficial effects on visual functions-such as best corrected visual acuity (BCVA), visual field (VF), multifocal electroretinography (mfERG), and microperimetry (MP)-in RP patients with various degrees of narrowed visual fields.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older;

* Diagnosis of any phenotypic variation of RP, confirmed by clinical history, fundus appearance, VF, and electroretinogram;
* Experience of various degrees of VF loss;
* BCVA from light perception of up to 110 letters (equal to 1.6 decimal values) in early treatment of diabetic retinopathy study (ETDRS) chart testing (Topcon CC-100 XP, Japan); & Mean deviation (MD) values from-33.0 to-5.0 dB with Humphrey or Octopus 900 visual field analysis (threshold 30-2, Sita Standard, Stimulus 3-white);
* Intraocular pressure (IOP) <22 mmHg.

Exclusion Criteria:

* The presence of cataracts or other media opacity that might affect the VF, MP, or mfERG recordings;

  * The presence of glaucoma, which causes visual field and optic disc changes;
  * The presence of any systemic disorder(e.g.,diabetes,neurological disease, or uncontrolled systemic hypertension) that may affect visual functions;
  * The habit of smoking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Visual field sensitivity | Change from baseline visual field sensitivity at 1 month
  A Humphrey or Octopus 900 visual field analyzer, threshold 30-2 modality, was used at time points of 0,1,2,and 3.In addition, it was used three times before application during experimentation to exclude the learning effect. The MD values, which were obtained from the baseline test and the final examination, were analyzed and compared statistically to make conclusions regarding effectiveness. Visual field analysis could be properly performed on patients whose BCVA values were better than 50 letters in ETDRS chart testing (0.1 decimal)

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent
Locations (1):
- Ankara University Biotechnology Institute, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koenekoop RK. Why some photoreceptors die, while others remain dormant: lessons from RPE65 and LRAT associated retinal dystrophies. Ophthalmic Genet. 2011 Jun;32(2):126-8. doi: 10.3109/13816810.2010.544361. Epub 2011 Jan 26. PMID 21268677
- [Background] Daftarian N, Kiani S, Zahabi A. Regenerative therapy for retinal disorders. J Ophthalmic Vis Res. 2010 Oct;5(4):250-64. PMID 22737370
- [Background] Anitua E, Muruzabal F, Tayebba A, Riestra A, Perez VL, Merayo-Lloves J, Orive G. Autologous serum and plasma rich in growth factors in ophthalmology: preclinical and clinical studies. Acta Ophthalmol. 2015 Dec;93(8):e605-14. doi: 10.1111/aos.12710. Epub 2015 Apr 2. PMID 25832910
- [Result] Arslan U, Ozmert E, Demirel S, Ornek F, Sermet F. Effects of subtenon-injected autologous platelet-rich plasma on visual functions in eyes with retinitis pigmentosa: preliminary clinical results. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):893-908. doi: 10.1007/s00417-018-3953-5. Epub 2018 Mar 15. PMID 29546474